CLINICAL TRIAL: NCT05865405
Title: Care Technology to Ascertain, Treat, and Engage the Community to Heal Depression in Patients With Multiple Sclerosis: Closing the Gaps in Depression Care for People With MS By Closing the Information Loop
Brief Title: A Closed Loop, Doctor to Patient, Mobile Application for Depression in People With Multiple Sclerosis
Acronym: MS-CATCH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 22-36620
Record Dates: First submitted 2023-04-24; First posted 2023-05-18 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis; MS; Depression
Keywords: MS; Multiple Sclerosis; Depression; Depressed
MeSH Terms: conditions — Multiple Sclerosis; Depression; Consciousness Disorders

STUDY DESIGN:
Intervention Model Description: Both arm 1 and arm 2 groups of participants will receive at least 6 months of MS CATCH tool intervention, with arm 1 receiving 12 months of intervention
Who Masked: Outcomes Assessor
Masking Description: The statistician will be blinded to what arm participants are a part of.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: 12 month MS CATCH tool intervention (Experimental): Participants in arm 1 will receive 12 months of use of the MS CATCH tool. This will include in-visit interventions and monthly questionnaires.
  Interventions: Behavioral: MS CATCH
- Arm 2: 6 month "usual care", 6 month MS CATCH tool intervention (Other): Participants in arm 2 will receive 6 months "usual care" followed by 6 months of MS CATCH tool intervention. These first 6 months will be used to assess the definition of "usual care".
  Interventions: Behavioral: MS CATCH

INTERVENTIONS:
Behavioral: MS CATCH — Participants will respond to a set of surveys every month to increase communication on mood with their clinician.

SUMMARY:
The researchers want to find out if an electronic application called MS CATCH can enhance patients' and doctors' experiences during and in between clinical visits. MS CATCH is a smartphone-based tool which allows patients to enter their mood related symptoms at regular intervals, which is then available to their Neurologist in their electronic medical record. The neurologist is also able to view additional information from their medical record, and receives alerts for changes reported by the patient that raise concern for the patient's mental health.

DETAILED DESCRIPTION:
MS-CATCH (Care technology to Ascertain, Treat, and engage the Community to Heal depression in patients with Multiple Sclerosis) is a behaviorally informed, digital health, closed-loop-intervention that brings longitudinal mood reporting into the point of care. It consists of a simple tool used by the patient to improve mood reporting. This then triggers real-time alerts delivered to the clinician, who can access a comprehensive dashboard featuring risk factors and interventions to be considered, as well as resources local to the patient. This dashboard launches straight from the patient's electronic health record (EHR). MS-CATCH was designed using extensive human-centered design in all phases of development, and HIPAA compliant REDCap for electronic data capture. While the tool requires institutional approvals to launch within the UCSF EHR, the design elements could be readily repurposed using these technologies to support other institutions' requirements. Each individual care component and visualization was then developed and refined using extensive stakeholder engagement and an eye to the COM-B (Capability, Opportunity, and Motivation to change Behavior) principles of behavioral change, in order to promote behaviors likely to improve depression reporting, screening, comprehensive treatment and follow through.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS (relapsing or progressive) by 2017 McDonald Criteria18
* Ages 18 to 80
* PHQ-9 score of 5-19
* Any MS therapy, or no treatment
* California resident to enable clinical telemedicine visits if warranted during the study visit

Exclusion Criteria:

* Cognitive dexterity or visual impairment (typically defined as corrected acuity less than 20/70) that, in the opinion of the study neurologist (RB), would put the participant at risk or limit their ability to adhere to the study protocol
* Inability to provide informed consent
* Psychotic disorders: bipolar disorder, schizophrenia, schizoaffective disorder
* Substance abuse that in the treating neurologist's perspective could influence the patient's safety on study or adherence to study protocol
* Another co-morbid CNS diagnosis eg. TBI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Mood Screening - Primary | 0-6 months, 0-12 months
  Clinician screening of depression as documented in the electronic health record (EHR)
Mood Reporting - Secondary | 6 months, Baseline, 12 months
  The percentage of patients who self-report mood at each clinical visit
Comprehensive Mood Evaluation - Secondary | 0-6 months, 0-12 months
  The percentage of depression risk factors evaluated at each clinical visit
Treatment recommendations - Secondary | 0-6 months, 0-12 months
  The percentage of visits in which applicable care was recommended; number of preventative care recommendations
Treatment recommendation follow-through - Secondary | 0-6 months, 0-12 months
  The number/percent of preventative care recommendations followed through by next visit
Adoption (uptake) - Primary | Initial month
  The percentage of patients using the tool during the first month of the study
Adoption (uptake) - Secondary | Baseline, 6 months
  The percentage of patient-clinician dyads who use the in-clinic dashboard at first visit

SECONDARY OUTCOMES:
Mood scores - Primary | Baseline, 3, 6, 9, and 12 months
  Hospital Anxiety Depression Scale (HADS) will be measured at baseline, 3, 6, 9, and 12 months, scale: 0-21 range for depressive scale, and 0-21 range for anxiety scale, with higher score meaning more depressive or anxious symptoms
Mood scores - Exploratory | 12 months
  Mini-International Neuropsychiatric Interview (MINI) assessment
Mood scores - Exploratory | 0-12 months, 0-6 months, 6-12 months
  Changes in Patient Health Questionnaire - 9 (PHQ-9), scale: 0-27, higher indicates more severe depressive symptoms
Other self-reported outcome - Modified Fatigue Impact Scale - Exploratory | 0-12 months, 0-6 months, 6-12 months
  Evaluating possible contributors to mood: fatigue (MFIS), scale: 0-84, higher score indicates more impact
Other self-reported outcome - Pittsburgh Sleep Quality Index - Exploratory | 0-12 months, 0-6 months, 6-12 months
  Evaluating possible contributors to mood: sleep (PSQI), scale: 0-21, higher scores indicates worse sleep quality
Other self-reported outcome - Oxford-Participation and Activities Questionnaire - Exploratory | 0-12 months, 0-6 months, 6-12 months
  Evaluating possible contributors to mood: engagement (Ox-PAQ), scale: 0-100, higher score indicates more problems with activity and participation
Other self-reported outcome - Impact on Participation and Autonomy - Exploratory | 0-12 months, 0-6 months, 6-12 months
  Evaluating possible contributors to mood: participation (IPA), scale: 0-128, with higher score indicating more impact on a person's autonomy and participation
Engagment (Sustained use) - Secondary | Every 3 months
  The percentage of patients who continue to use the patient-facing tool at least quarterly
Engagement (Sustained use) - Secondary | 12 months
  The percentage of patient-clinician dyads in Arm 1 (early start) who continued to use the tool at the 12 month visit
Engagement (Sustained use) - Exploratory | Baseline, 6 month, 12 month
  Length of each session
Engagement (Sustained use) - Exploratoy | 12 month
  Qualitative feedback in exit interviews
Engagement (Sustained use) - Exploratory | 12 month
  Net promoter score (NPS)
Adherence - Secondary | 12 months
  The percentage of depression-reporting prompts responded to per participant on their patient-facing tool; the percentage participants responding to >75% depression prompts

OTHER OUTCOMES:
Trial retention - Exploratory | 12 months
  Trial retention
Self-Efficacy - Exploratory | Baseline-12 months
  Changes in patient reported self efficacy at managing a chronic disease, reported using the "Self-efficacy for Managing a Chronic Disease 6-item Scale" (Lorig) Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Riley Bove, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Weill Institute for Neurosciences, University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The deidentified dataset will be shared with qualified collaborators upon request, provision of CITI and other certifications, and data sharing agreement. We will share the results, once the data are complete and analyzed, with the scientific community and patient/clinician participants through abstracts, presentations and manuscripts.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months post trial
Access Criteria: Qualified collaborators upon request, provision of CITI and other certifications, and data sharing agreement

REFERENCES:
- [Derived] Henderson K, Reihm J, Koshal K, Wijangco J, Sara N, Miller N, Doyle M, Mallory A, Sheridan J, Guo CY, Oommen L, Rankin KP, Sanders S, Feinstein A, Mangurian C, Bove R. A Closed-Loop Digital Health Tool to Improve Depression Care in Multiple Sclerosis: Iterative Design and Cross-Sectional Pilot Randomized Controlled Trial and its Impact on Depression Care. JMIR Form Res. 2024 Mar 15;8:e52809. doi: 10.2196/52809. PMID 38488827
- [Derived] Henderson K, Reihm J, Koshal K, Wijangco J, Miller N, Sara N, Doyle M, Mallory A, Sheridan J, Guo CY, Oommen L, Feinstein A, Mangurian C, Lazar A, Bove R. Pragmatic phase II clinical trial to improve depression care in a real-world diverse MS cohort from an academic MS centre in Northern California: MS CATCH study protocol. BMJ Open. 2024 Feb 24;14(2):e077432. doi: 10.1136/bmjopen-2023-077432. PMID 38401894